CLINICAL TRIAL: NCT06203340
Title: Investigation of the Effectiveness of Lumbar Training or Core Stabilisation Exercises on Pain, Mobilisation and Quality of Life in Patients with Chronic Low Back Pain: a Randomised Controlled Study
Brief Title: Lumbar School Training or Core Stabilization Exercises on Pain, Mobilization and Quality of Life Low Back Pain
Acronym: Lowbackpain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, MUSA ÇANKAYA, Lecturer Doctor, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MUSACANKAYA
Record Dates: First submitted 2023-12-27; First posted 2024-01-12 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Low Back Pain; Core Stability; Core-based Exercise; Back School
Keywords: Back schools; Low back pain; Exercise; Physical therapy
MeSH Terms: conditions — Low Back Pain; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Posttest and control grouped randomized controlled clinical trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Lumbar school training (Experimental): Lumbar back school is a programme for patient groups that provides information about the anatomy, biomechanics, optimal posture, ergonomics and lumbar exercises.
  The aim of the lumbar lumbar school school is to reduce low back pain and to teach the individual to take care of his lumbar. It is applied to increase the skills of individuals to solve the problems they encounter in daily life and to teach them ways of coping. Assessment of the patient, explanation of the anatomy, functions and pathophysiology of low back pain, appropriate posture, use of correct body mechanics and theoretical explanation of exercise.
  Interventions: Other: Core stabilizasyon and lumbal back school
- Core stabilisation training (Experimental): Core exercise programmes are designed to improve stabilisation, strength and power. Core exercise programmes are aimed to improve the sense of bodily movement and position (proprioception), which systematically progresses, prepares for activities and goals. Patients are started from the beginning level of the core exercises and in the following weeks, to the extent that the patients can do will be made more difficult.
  Interventions: Other: Core stabilizasyon and lumbal back school
- Control group (No Intervention): Patients with a previous diagnosis of pain in the lumbar region will be sought. Patients will be invited to the institution and will be informed about low back pain. Patients with low back pain will be evaluated with self-report scales and functional tests. No treatment will be applied as a treatment.

INTERVENTIONS:
Other: Core stabilizasyon and lumbal back school — Lumbal back schooL
  Other Names: Exercise training:
  Arms: Core stabilisation training; Lumbar school training

SUMMARY:
Chronic low back pain (CLBP) is defined as low back pain lasting longer than three months. CLBP is one of the most common and expensive diseases in terms of both labour loss and treatment costs, and it is very important to treat it with conventional (non-surgical) treatment methods. Clinical guidelines recommend active treatments that address psychosocial factors and focus on functional improvement. Within this approach, low back protection training, called low back school, is recognised as an effective and economical method. This study was planned to investigate the effectiveness of lumbar school training or core stabilisation exercises on pain, mobilisation and quality of life in patients with chronic low back pain.

In this research, patients coming to Seydişehir State Hospital physiotherapy unit will be included in the study. Patients will be taken in Seydişehir Vocational School of Health Services Vocational School vocational skills laboratory and Seydişehir State Hospital physiotherapy unit. As a result of the power analysis, 64 patients are planned to be included. Simple randomisation will be used. Sealed opaque envelopes will be prepared by the research team. Opaque envelopes will be determined as 24 (core exercise group) and 24 (B) (lumbar school), 24 C kontrol. The pain intensity of the patients will be determined by the Visual Analogue Scale, which is a self-report scale, and the functional disability levels will be determined by the Oswestry Disability Index and the quality of life levels will be determined by the World Health Organization Quality of Life Module (WHOQOL-BREF) and spinal mobility will be determined by measuring the hand-finger ground distance.

Patients will be divided into two groups as core exercise group and lumbar school training group and will be evaluated before and after treatment and training.

Keywords: Chronic low back pain, back school, core stabilisation exercise

DETAILED DESCRIPTION:
Low back pain is defined as pain, increased muscle tension or stiffness localised between the costal margin and lower gluteal folds and associated with lower extremity pain (1).

Between 70-85% of people experience low back pain throughout their lives. Almost 20% of these cases become permanent (2). Chronic low back pain (CLBP) is defined as low back pain lasting longer than three months. It is a worldwide common disease that imposes a significant medical and economic burden on individuals and society (3). Mechanical low back pain is defined as a clinical picture that develops as a result of overuse, strain or traumatisation or deformation of the structures forming the spine. In order to define low back pain as mechanical, all organic causes such as inflammatory, infectious, tumoural, metabolic causes, fractures and pain reflected from internal organs should be excluded (4).

It is very important that CLBP, which is very common in the society and is one of the most expensive diseases in terms of both labour loss and treatment cost, is treated with conventional (non-surgical) treatment methods (7). It has been reported that medical, psychological, physical approaches and multidisciplinary methods are effective in the treatment of CLBP(13). In the last thirty years, changes have been made in the basic recommendations in clinical practice guidelines. Self-management, physical, psychological therapies and some complementary medicine treatments are now given more importance and pharmacological and surgical treatments are less preferred. Guidelines recommend active treatments that address psychosocial factors and focus on functional recovery (14). Within this approach, waist protection training, which is called waist school, is accepted as an effective and economical method (5).

The lumbar school method was developed by Mariane Zachrisson Forssel in Sweden in 1969 with the aim of managing the patient's current condition and preventing recurrent low back pain (6). The programme consists of 4 sessions lasting approximately 45 minutes and each session is organised with theoretical components and includes exercises to improve mobility (5). Standard training strategies can be used in patients with chronic low back pain. However, it is not sufficient as a treatment alone. Standard training strategies should include exercise-related practices (7). Clinical guidelines state that trunk coordination, strengthening and endurance exercises should be utilised to reduce the disability in CLBP (7,8). Various therapeutic exercises are applied in clinical practice for CBLP patients.

Core stabilisation exercises (CSE) are based on a motor learning approach and provide the activation of the transversus abdominis and lumbar multifidus muscles together. These deep stabilisation muscles increase intra-abdominal pressure by adhering to the thoraco-lumbar fascia. It has a firming effect on the lumbar spine. It increases the segmental stability of the spine (9). In addition, CSE reduces pain by reversing the pain-related structuring in the motor cortex. It improves muscle strength and improves neuromuscular control of spinal stability. CSE increases the sense of proprioception and successfully corrects postural disorders (10).

Although many different interventions are widely used in physiotherapy clinics, there are few studies evaluating the effects of lumbar school and CSE, and no studies comparing their effectiveness with each other have been found. Therefore, the aim of the present study was to investigate the comparative efficacy of lumbar school training or core stabilisation exercises on pain, mobilisation and quality of life in patients with CBLP.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 55,
* Having low back pain for at least 3 months (12 hf),
* Score 14% or more on the Oswestry Disability Index,
* Ability to move independently (with or without assistance), to participate in a rehabilitation program and to read, write and understand Turkish well enough to complete questionnaires independently.

Exclusion Criteria:

* VAS score < 20 mm),
* Those with cognitive impairment that prevents them from understanding and completing the questionnaire,
* Aphasic patients, patients unwilling to volunteer, patients with specific etiology of low back pain such as inflammatory, infectious, tumoral, fracture and visceral pain.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2024-01-02 (Actual); Primary Completion 2024-05-05 (Actual); Study Completion 2024-09-07 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | Evaluation will be made before and after treatment. The evaluation is expected to take 20 minutes in total.
  It is a scale that assesses the severity of pain and consists of a single 10-centimeter line. Patients will be asked to mark the intensity of their pain at rest, during activity (movement) and at night on two separate 10-centimeter lines. The starting point on the scale is defined as no pain and the end point is defined as the most severe unbearable pain. During the calculation, the distance between the marked point and the starting point is measured in centimeters. The relationship of pain intensity with activity (VAS-movement, VAS-rest) and night pain (VAS-night) will be questioned separately. An increase in the score means an increase in pain intensity.
Oswestry Disability Index | Evaluation will be made before and after treatment. The evaluation is expected to take 20 minutes in total.
  It was developed to evaluate the degree of loss of function in low back pain. The Oswestry Disability Index, whose validity and reliability in Turkish was demonstrated in 2004, consists of 10 items. Items question pain severity, self-care, lifting and carrying, walking, sitting, standing, sleep, degree of pain change, travel and social life. Under each item there are six statements in which the patient ticks the one appropriate to his/her situation. The first statement is scored as "0" and the sixth statement is scored as "5". When the total score is calculated, it is multiplied by two and expressed as a percentage. The maximum score is "100" and the minimum score is "0". As the total score increases, the disability level also increases.
World Health Organization Quality of Life Module (WHOQOL-BREF) | Evaluation will be made before and after treatment. The evaluation is expected to take 20 minutes in total.
  WHOQOL, a general-purpose quality of life profile scale, has two versions: long and short. The health-related quality of life scale was developed by WHO and its validity and reliability were tested by Eser et al. The scale has two versions: long (WHOQOL-100) and short (WHOQOL-27) form. The scale measures physical, spiritual, social and environmental well-being and consists of 26 questions. The scale can be applied to non-elderly adults. The scale was also applied to healthcare workers. Since each domain expresses the quality of life in its own field independently of each other, domain scores are calculated between 4-20. As the score increases, the quality of life increases.
Lumbar flexion (Hand-finger ground distance) | Evaluation will be made before and after treatment. The evaluation is expected to take 20 minutes in total.
  HFGD, the patient was asked to stand in an upright posture on a horizontal straight line with a distance of 30 cm between both medial malleolus and to evaluate his hands on the ground without bending his knees. The distance between the middle finger and the floor will be measured.
  It will also be evaluated with an inclinometer. It was developed by Mayer et al. This technique, recommended by the American Medical Association, is a non-invasive and easy-to-apply method. The advantages of the method are its low cost, ability to evaluate pelvic and lumbar spine movements separately, and easy applicability. Its validity and reliability have been demonstrated by many studies.
Lumbar lateral flexion | Evaluation will be made before and after treatment. The evaluation is expected to take 20 minutes in total.
  The distance between the fingertip and the ground will be measured while the patient is standing, then he will be asked to lean to the right side and the distance between the ground and the fingertip will be measured again. The same process will be repeated for the left side and the average of the measurements of the right and left sides will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Havva CİNGÖZ, M.Dr., Study Chair — Seydişehir Devlet Hastanesi (Seydişehir/KONYA; Musa Çankaya, Pt. PhD, Study Director — Necmettin Erbakan University
Locations (1):
- Musa Çankaya, Konya, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ozsoy G, Ilcin N, Ozsoy I, Gurpinar B, Buyukturan O, Buyukturan B, Kararti C, Sas S. The Effects Of Myofascial Release Technique Combined With Core Stabilization Exercise In Elderly With Non-Specific Low Back Pain: A Randomized Controlled, Single-Blind Study. Clin Interv Aging. 2019 Oct 9;14:1729-1740. doi: 10.2147/CIA.S223905. eCollection 2019. PMID 31631992
- [Background] Ghaderi Niri H, Ghanavati T, Mostafaee N, Salahzadeh Z, Divandari A, Adigozali H, Ahadi J. Oswestry Disability Index, Roland-Morris Disability Questionnaire, and Quebec Back Pain Disability Scale: Responsiveness and Minimal Clinically Important Changes in Iranian People with Lumbar Disc Herniation Following Physiotherapy. Arch Bone Jt Surg. 2024;12(1):58-65. doi: 10.22038/ABJS.2023.72246.3366. PMID 38318303
- [Background] Alqhtani RS, Ahmed H, Ghulam HSH, Alyami AM, Al Sharyah YHH, Ahmed R, Khan A, Khan AR. Efficacy of Core-Strengthening and Intensive Dynamic Back Exercises on Pain, Core Muscle Endurance, and Functional Disability in Patients with Chronic Non-Specific Low Back Pain: A Randomized Comparative Study. J Clin Med. 2024 Jan 15;13(2):475. doi: 10.3390/jcm13020475. PMID 38256609
- [Background] Jenks A, Hoekstra T, van Tulder M, Ostelo RW, Rubinstein SM, Chiarotto A. Roland-Morris Disability Questionnaire, Oswestry Disability Index, and Quebec Back Pain Disability Scale: Which Has Superior Measurement Properties in Older Adults With Low Back Pain? J Orthop Sports Phys Ther. 2022 Jul;52(7):457-469. doi: 10.2519/jospt.2022.10802. Epub 2022 May 18. PMID 35584027
- [Background] Rajfur J, Rajfur K, Kosowski L, Walewicz K, Dymarek R, Ptaszkowski K, Taradaj J. The effectiveness of dry needling in patients with chronic low back pain: a prospective, randomized, single-blinded study. Sci Rep. 2022 Sep 22;12(1):15803. doi: 10.1038/s41598-022-19980-1. PMID 36138055
- [Background] Kleine-Borgmann J, Dietz TN, Schmidt K, Bingel U. No long-term effects after a 3-week open-label placebo treatment for chronic low back pain: a 3-year follow-up of a randomized controlled trial. Pain. 2023 Mar 1;164(3):645-652. doi: 10.1097/j.pain.0000000000002752. Epub 2022 Aug 10. PMID 35947884
- [Background] Lara-Palomo IC, Gil-Martinez E, Antequera-Soler E, Castro-Sanchez AM, Fernandez-Sanchez M, Garcia-Lopez H. Electrical dry needling versus conventional physiotherapy in the treatment of active and latent myofascial trigger points in patients with nonspecific chronic low back pain. Trials. 2022 Mar 28;23(1):238. doi: 10.1186/s13063-022-06179-y. PMID 35346331
- [Background] Kim B, Yim J. Core Stability and Hip Exercises Improve Physical Function and Activity in Patients with Non-Specific Low Back Pain: A Randomized Controlled Trial. Tohoku J Exp Med. 2020 Jul;251(3):193-206. doi: 10.1620/tjem.251.193. PMID 32669487
- [Background] Minghelli B, Nunes C, Oliveira R. Back School Postural Education Program: Comparison of Two Types of Interventions in Improving Ergonomic Knowledge about Postures and Reducing Low Back Pain in Adolescents. Int J Environ Res Public Health. 2021 Apr 22;18(9):4434. doi: 10.3390/ijerph18094434. PMID 33921952
- [Background] Ahmadi H, Adib H, Selk-Ghaffari M, Shafizad M, Moradi S, Madani Z, Partovi G, Mahmoodi A. Comparison of the effects of the Feldenkrais method versus core stability exercise in the management of chronic low back pain: a randomised control trial. Clin Rehabil. 2020 Dec;34(12):1449-1457. doi: 10.1177/0269215520947069. Epub 2020 Jul 29. PMID 32723088
- [Background] Hajihasani A, Rouhani M, Salavati M, Hedayati R, Kahlaee AH. The Influence of Cognitive Behavioral Therapy on Pain, Quality of Life, and Depression in Patients Receiving Physical Therapy for Chronic Low Back Pain: A Systematic Review. PM R. 2019 Feb;11(2):167-176. doi: 10.1016/j.pmrj.2018.09.029. Epub 2019 Feb 11. PMID 30266349